CLINICAL TRIAL: NCT00578214
Title: Randomized Controlled and Prospective Studies of Safety and Efficacy of Oral Midazolam for Perioperative Anxiolysis of Patients Undergoing Mohs Micrographic Surgery.
Brief Title: Safety and Efficacy of Oral Midazolam for Perioperative Anxiety Relief of Patients Undergoing Mohs Micrographic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Larisa Ravitskiy, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-000848
Record Dates: First submitted 2007-12-20; First posted 2007-12-21 (Estimated); Results first posted 2012-02-09 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Basal Cell Carcinoma; Squamous Cell Carcinoma; Skin Cancer; Anxiety
Keywords: mohs micrographic surgery; skin cancer; anxiety; basal cell carcinoma; squamous cell carcinoma; midazolam; versed
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Skin Neoplasms; Anxiety Disorders | interventions — Midazolam; Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Randomized Midazolam (Active Comparator): Single-dose midazolam
  Interventions: Drug: Randomized Midazolam; Drug: Local Anesthesia
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo; Drug: Local Anesthesia
- Prospective Midazolam (Experimental)
  Interventions: Drug: Local Anesthesia; Drug: Prospective Midazolam

INTERVENTIONS:
Drug: Randomized Midazolam — Midazolam was prepared in a 2 mg/ml cherry flavored syrup. In the randomized arm, patients received a single-dose administration of 5 ml (10 mg) of the midazolam syrup.
  Other Names: Versed
  Arms: Randomized Midazolam
Other: Placebo — The placebo was prepared as a color- and texture-matched cherry flavored syrup without midazolam.
  Arms: Placebo
Drug: Local Anesthesia — Lidocaine 1% with 1:100,000 epinephrine
Drug: Prospective Midazolam — Midazolam was prepared in a 2 mg/ml cherry flavored syrup. Dosing in the prospective arm was based on weight (>45 to 77 kg, 10 mg; >77 to 100 kg, 15 mg; greater than or equal to 100 kg, 20 mg). In the prospective arm patients were given additional doses of midazolam as necessary (in 5 mg increments) to achieve and maintain the desired level of anxiolysis.
  Other Names: Versed
  Arms: Prospective Midazolam

SUMMARY:
Midazolam is an approved sedative medication used for medical procedures. This study was being done to document the safety and efficacy of midazolam in improving anxiety, heart rate, and blood pressure in patients prior to undergoing Mohs micrographic surgery for the treatment of skin cancer (basal cell carcinoma or squamous cell carcinoma). Midazolam may make a patient relaxed and sleepy, and lower blood pressure. These effects last for about 2 hours.

This study had two parts. In the first part, eligible patients were randomized to either receiving one standard dose of midazolam syrup or placebo syrup before their surgery, with neither the patient nor the study team knowing which patient received the study drug. In the second part, patients who were not eligible to participate in the randomized study or who refused to participate in the randomized study were enrolled in a prospective arm where they knew they were receiving midazolam syrup. In the prospective arm, the doses were based on the patient's weight, and patients were given additional doses of midazolam syrup as necessary to control their anxiety.

The primary hypothesis of this study was that a single dose of oral midazolam syrup to patients prior undergoing outpatient Mohs micrographic surgery for skin cancer would result in lower anxiety scores at 60 minutes compared to placebo. In addition, the second hypothesis of this study was that patients given oral midazolam would have the rate of adverse events that was not worse than 25% higher than in the placebo group.

DETAILED DESCRIPTION:
The main objective of this study was to establish the safety and efficacy of midazolam in patients with skin cancer undergoing outpatient Mohs micrographic surgery. Patients were randomized in a double-blind placebo-controlled study of a single-dose midazolam syrup for efficacy in producing safe anxiolysis of short duration. A parallel prospective arm of the study involved administration of midazolam in an unblinded fashion. Based on available studies of orally administered midazolam, the expectation was that the only observed adverse events will be minor and the major adverse event rate for midazolam would be similar to placebo. Data was collected on vital signs, anxiety, adverse events, and overall satisfaction with the anxiolytic agent.

ELIGIBILITY:
Inclusion Criteria:

- 1 or 2 sites of biopsy-confirmed squamous cell or basal cell carcinomas limited to head and neck regions

Inclusion Criteria for Prospective Arm:

* Patients wishing to receive oral midazolam in a non-blinded fashion will not be excluded based on the size of an individual tumor, total number of tumors, or prior history of oral midazolam
* No upper weight limitation

Exclusion Criteria:

* Prior history of allergy to midazolam or any of the syrup components
* History of hypersensitivity to other benzodiazepines
* Congestive heart failure (AHA Class III and IV)
* Renal failure requiring hemodialysis
* End-stage liver failure
* Chronic alcoholism or alcohol intoxication within 24 hours of surgery
* Untreated or uncontrolled open angle glaucoma
* Uncontrolled hypertension
* History of psychoses or affective disorders
* Neuromuscular disorders such as myasthenia gravis
* Chronic obstructive pulmonary disease
* Patients on medications interfering with renal excretion or microsomal metabolism unless the last dose was taken greater than or equal to 5 half-lives prior to surgery
* Patients weighing less than 100 lb (45 kg)
* Pregnant women; women of childbearing potential will be required to take an in-office urine pregnancy test.
* Breast-feeding mothers must stop breast-feeding for 7 days after taking midazolam to take part in this study

Additional Exclusion Criteria for Randomized Arms:

* Patients with a single cancer > 5 cm in the greatest dimension or with more than 2 cancers
* Patients who were previously premedicated with oral midazolam during prior Mohs micrographic surgery episodes
* Patients weighing more than 220 lb (100 kg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-03; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clark C Otley, MD, Principal Investigator — Mayo Clinic; Larisa Ravitskiy, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Ravitskiy L, Phillips PK, Roenigk RK, Weaver AL, Killian JM, Hoverson Schott A, Otley CC. The use of oral midazolam for perioperative anxiolysis of healthy patients undergoing Mohs surgery: conclusions from randomized controlled and prospective studies. J Am Acad Dermatol. 2011 Feb;64(2):310-22. doi: 10.1016/j.jaad.2010.02.038. PMID 21238825

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing outpatient Mohs surgery at the Mayo Clinic in Rochester, MN were included in either the randomized arms (midazolam vs placebo) or in the prospective midazolam arm. The study was performed between March 2007 and June 2008.
Groups:
- Randomized Midazolam: Randomized patients receiving single-dose midazolam syrup
- Placebo: Randomized patients receiving placebo syrup
- Prospective Midazolam: Open-label, dose of Midazolam based on patient's weight, additional doses to control anxiety were possible
Period: Overall Study
Arm/Group | Randomized Midazolam | Placebo | Prospective Midazolam
Started | 22 | 22 | 31
Completed | 22 | 22 | 31
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized Midazolam | Placebo | Prospective Midazolam | Total
Number analyzed (Participants) | 22 | 22 | 31 | 75
Age Continuous [Mean (Standard Deviation); unit: years] | 71.9 (11.5) | 70.1 (12.8) | 62.9 (14.1) | 67.7 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 21 | 40
  Male | 13 | 12 | 10 | 35
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 31 | 75
Weight at study entry [Mean (Standard Deviation); unit: kg] | 83.1 (13.23) | 80.6 (11.82) | 87.8 (20.16) | 84.3 (16.2)
Prior Mohs Micrographic Surgery [Number; unit: participants]
  No | 16 | 17 | 21 | 54
  Yes | 5 | 4 | 9 | 18
  Unknown | 1 | 1 | 1 | 3
Type of Non-melanoma Skin Cancer [Number; unit: participants]
  Basal Cell Carcinoma | 13 | 11 | 22 | 46
  Squamous Cell Carcinoma | 9 | 10 | 8 | 27
  Basal Cell and Squamous Cell Carcinomas | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Patient Anxiety at Baseline
Description: A 10-point visual analog scale (VAS) was used to measure anxiety. The patients marked on the scale their feeling of anxiety. The lowest value possible was 0 (no anxiety) and the highest value possible was 10 (highest possible anxiety).
Time Frame: Baseline (prior to drug administration)
Population: The analysis was done on the patients who completed the assessment. One patient in the randomized midazolam arm, 2 patients in the placebo arm, and 1 patient in the prospective midazolam arm did not complete this assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Midazolam | Placebo | Prospective Midazolam
Number analyzed (Participants) | 21 | 20 | 30
units on a scale | 1.3 (1.5) | 1.4 (1.6) | 3.4 (2.7)

2. Secondary Outcome: Patient Alertness at Baseline
Description: A 10-point visual analog scale (VAS) was used to measure alertness. The patients marked on the scale their feeling of alertness. The lowest value possible was 0 (awake) and the highest value possible was 10 (barely awake).
Time Frame: Baseline (prior to drug administration)
Population: The analysis was done on the patients who completed the assessment. One patient in the randomized midazolam arm did not complete this assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Midazolam | Placebo | Prospective Midazolam
Number analyzed (Participants) | 21 | 22 | 31
units on a scale | 0.2 (0.6) | 0.2 (0.7) | 0.2 (0.6)

3. Secondary Outcome: Patient Alertness at 60 and 120 Minutes
Description: as for outcome 2
Time Frame: 60 and 120 minutes after drug administration
Population: The analysis was done on the patients who completed the assessment. One patient in the randomized midazolam arm and 1 patient in the prospective midazolam arm did not complete this assessment.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Randomized Midazolam | Placebo | Prospective Midazolam
Number analyzed (Participants) | 21 | 22 | 30
units on a scale
  60 min patient alertness | 3.7 (4.0) | 0.7 (1.6) | 5.1 (3.4)
  120 min patient alertness | 2.1 (2.9) | 0.5 (1.1) | 3.4 (2.9)

4. Primary Outcome: Patient Anxiety at 60 and 120 Minutes
Description: as for outcome 1
Time Frame: 60 and 120 minutes after drug administration
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Midazolam | Placebo | Prospective Midazolam
Number analyzed (Participants) | 21 | 22 | 31
units on a scale
  60 min patient anxiety | 0.1 (0.5) | 0.8 (0.9) | 1.0 (1.7)
  120 min patient anxiety | 0.2 (0.5) | 0.4 (0.8) | 0.8 (1.6)

5. Secondary Outcome: Patient Cognitive Function at Baseline and 60 Minutes
Description: Cognitive function was measured by the Mini-Mental State Examination (MMSE), a brief 30 point questionnaire test. The scores can range from 0 (low cognitive function) to 30 (high cognitive function).
Time Frame: baseline (prior to drug administration) and 60 minutes after drug administration
Population: The analysis was done on the patients who completed the assessment. One patient in the prospective midazolam arm did not complete this assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Midazolam | Placebo | Prospective Midazolam
Number analyzed (Participants) | 22 | 22 | 30
units on a scale
  Baseline Cognitive Function | 28.9 (1.4) | 29.3 (0.9) | 29.2 (1.9)
  60 min Cognitive Function | 22.9 (10.6) | 29.4 (0.7) | 24.3 (10.9)

6. Secondary Outcome: Patient Cognitive Function at 120 Minutes
Description: as for outcome 5
Time Frame: 120 minutes after drug administration
Population: The analysis was done on the patients who completed the assessment. Two patients in the placebo arm did not complete this assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Midazolam | Placebo | Prospective Midazolam
Number analyzed (Participants) | 22 | 20 | 31
units on a scale | 26.0 (8.6) | 29.2 (1.2) | 27.5 (7.0)

7. Secondary Outcome: Blood Pressure at 30 Minutes
Time Frame: 30 minutes after drug administration
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Randomized Midazolam | Placebo | Prospective Midazolam
Number analyzed (Participants) | 22 | 22 | 31
mm Hg
  30 min Systolic Blood Pressure | 121.4 (19.50) | 125.9 (12.24) | 118.5 (16.99)
  30 min Diastolic Blood Pressure | 67.1 (12.9) | 68.4 (7.82) | 63.2 (10.58)

8. Secondary Outcome: Heart Rate at 30 Minutes
Time Frame: 30 minutes after drug administration
Population: The analysis was done on the patients who completed the assessment. One patient in the placebo arm did not complete this assessment.
Measure: Mean (Standard Deviation); unit: heart beats per minute
Arm/Group | Randomized Midazolam | Placebo | Prospective Midazolam
Number analyzed (Participants) | 22 | 21 | 31
heart beats per minute | 61.7 (14.84) | 64.3 (8.16) | 72.1 (12.65)

9. Secondary Outcome: Respiratory Rate at 30 Minutes
Time Frame: 30 minutes after drug administration
Population: The analysis was done on the patients who completed the assessment. Three patients in the randomized midazolam arm and 2 patients in the placebo arm did not complete this assessment.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Randomized Midazolam | Placebo | Prospective Midazolam
Number analyzed (Participants) | 19 | 20 | 31
breaths per minute | 19.4 (12.26) | 16.1 (2.63) | 16.2 (3.07)

10. Secondary Outcome: Pulse Oximetry at 30 Minutes
Description: Pulse oximetry measures the oxygenation of a patient's hemoglobin. A sensor is placed on the patient's finger. Light at red and infrared wavelengths is passed sequentially through the patient to a photodetector. The changing absorbance at each of the two wavelengths is measured, allowing determination of the absorbance. The color of the blood provides a measure of oxygenation (the percentage of hemoglobin molecules bound with oxygen molecules). A healthy young person will probably have an oxygen saturation of 95-99%.
Time Frame: 30 minutes after drug administration
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage of oxygenation
Arm/Group | Randomized Midazolam | Placebo | Prospective Midazolam
Number analyzed (Participants) | 19 | 20 | 31
percentage of oxygenation | 94.5 (2.18) | 95.6 (2.11) | 95.6 (2.56)

11. Secondary Outcome: Blood Pressure at 60 Minutes
Time Frame: 60 minutes after drug administration
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Randomized Midazolam | Placebo | Prospective Midazolam
Number analyzed (Participants) | 19 | 20 | 31
mm Hg
  60 min systolic blood pressure | 120.1 (18.10) | 131.9 (14.59) | 113.5 (15.61)
  60 min diastolic blood pressure | 65.3 (9.17) | 69.5 (8.69) | 61.5 (10.04)

12. Secondary Outcome: Heart Rate at 60 Minutes
Time Frame: 60 minutes after drug administration
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: heart beats per minute
Arm/Group | Randomized Midazolam | Placebo | Prospective Midazolam
Number analyzed (Participants) | 19 | 20 | 31
heart beats per minute | 60.3 (13.94) | 61.4 (7.45) | 69.6 (10.75)

13. Secondary Outcome: Respiratory Rate at 60 Minutes
Time Frame: 60 minutes after drug administration
Population: The analysis was done on the patients who completed the assessment. Three patients in the randomized midazolam arm and 3 patients in the placebo arm did not complete this assessment.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Randomized Midazolam | Placebo | Prospective Midazolam
Number analyzed (Participants) | 19 | 19 | 31
breaths per minute | 20.6 (12.33) | 16.3 (2.43) | 16.8 (2.69)

14. Secondary Outcome: Pulse Oximetry at 60 Minutes
Description: as for outcome 10
Time Frame: 60 minutes after drug administration
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage of oxygenation
Arm/Group | Randomized Midazolam | Placebo | Prospective Midazolam
Number analyzed (Participants) | 19 | 19 | 31
percentage of oxygenation | 94.5 (2.43) | 96.4 (1.81) | 95.5 (3.03)

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events (AEs) during the 120 minutes after drug administration. Patients also were contacted by phone within 24 hours of the procedure using a specific inventory questionnaire to determine if there were any delayed AEs.
Arm/Group | Randomized Midazolam | Placebo | Prospective Midazolam
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/31
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 1/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Midazolam (N=22) | Placebo (N=22) | Prospective Midazolam (N=31)
Mild and transient hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was hindered by slow accrual and fell short of reaching the target number of patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No